CLINICAL TRIAL: NCT04268667
Title: A Comparative Study Between Cervicothoracic and Upper Cervical Spine Manipulation in Patients With Chronic Mechanical Neck Pain: a Randomized Controlled Trial
Brief Title: Comparison of Two Spinal Manipulation Treatments in Patients With Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica Ciudad de Almería (Other)
Responsible Party: Principal Investigator, Raúl Romero del Rey, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: spinal manipulation
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain
Keywords: disability evaluation; musculoskeletal manipulations; neck pain; spinal manipulation
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upper cervical spine manipulation group (Experimental): Spinal thrust joint manipulation on the atlantoaxial joint
  Interventions: Other: Spinal manipulation
- Cervicothoracic spine manipulations group (Active Comparator): Different spinal thrust joint manipulations on the thoracic spine (T6), mid-cervical spine (C3-C4) and cervicothoracic junction (C7-T1).
  Interventions: Other: Spinal manipulation

INTERVENTIONS:
Other: Spinal manipulation — Application of upper cervical spine thrust joint manipulation or application of a full combination of cervical, cervico-thoracic and thoracic spine thrust joint manipulation.

SUMMARY:
There is enough evidence to suggest that the spinal manipulation of the upper cervical spine and cervicothoracic spine are effective in decreasing neck pain. Therefore, the purpose of this randomized controlled trial is to compare the effects of an isolated application of upper cervical spine thrust joint manipulation with the application of a full combination of cervical, cervico-thoracic and thoracic spine thrust joint manipulation on neck pain, disability and cervical range of motion in individuals with chronic mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Symptom persistence for more than 12 weeks.
* Age from 18 to 55 years.
* Localized pain in the cervical spine.
* Symptoms are caused by cervical movement or sustained postures.

Exclusion Criteria:

* Stage acute of symptoms.
* Any contraindication to cervical spinal manipulation (fracture, osteoporosis, joint infections or vertebrobasilar insufficiency).
* Patients with previous neck trauma or cervical spine surgery.
* Patients diagnosed with cervical radiculopathy.
* Patients diagnosed with fibromyalgia.
* Have been treated with manual therapy in the last 3 months.
* Receiving other treatment during the course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Change in neck pain at rest: Numeric Pain Rating Scale (0-10) | Baseline and 7 days post-treatment
  Neck pain at rest. Measured with the Numeric Pain Rating Scale (0 = ''no pain'' and 10 = ''worst imaginable pain).
Change in neck disability: Neck Disability Index (0-50) | Baseline and 7 days post-treatment
  Neck disability is measured with Neck Disability Index (10 items). A higher score indicates greater disability.

SECONDARY OUTCOMES:
Change in flexion movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in flexion. Measured with a Cervical Range of Motion (CROM) device
Change in extension movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in extension. Measured with a Cervical Range of Motion (CROM) device
Change in rigth lateral flexion movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in right lateral flexion. Measured with a Cervical Range of Motion (CROM) device
Change in left lateral flexion movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in left lateral flexion. Measured with a Cervical Range of Motion (CROM) device
Change in right rotation movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in right rotation. Measured with a Cervical Range of Motion (CROM) device
Change in left rotation movement: Cervical Range of Motion device | Baseline and 7 days post-treatment
  Range of cervical motion in left rotation. Measured with a Cervical Range of Motion (CROM) device

CONTACTS AND LOCATIONS:
Overall Officials: Raúl Romero del Rey, Mr, Principal Investigator — Clinica Ciudad de Almería
Locations (1):
- Clínica Ciudad de Almería, Almería, Spain